CLINICAL TRIAL: NCT02135536
Title: A Phase 2, Multi-Center Study to Evaluate Three Doses of NGM282 Administered for 24 Weeks in Patients With Primary Biliary Cirrhosis (PBC) Who Have Completed Study 13-0103
Brief Title: Phase 2b Study of NGM282 Extended Treatment in Patients With Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Collaborators: NGM Biopharmaceuticals Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-0104
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NGM282 Dose 1 (Experimental): NGM282 Dose 1
  Interventions: Biological: NGM282
- NGM282 Dose 2 (Experimental): NGM282 Dose 2
  Interventions: Biological: NGM282
- NGM282 Dose 3 (Experimental): NGM282 Dose 3
  Interventions: Biological: NGM282

INTERVENTIONS:
Biological: NGM282 — NGM282

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and activity of extended treatment with NGM282 in patients with Primary Biliary Cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Completion of NGM 13-0103
* Males or females, between 18 and 75 years of age, inclusive
* PBC Diagnosis consistent with AASLD and EASL guidelines
* Stable dose of UDCA

Exclusion Criteria:

* Chronic liver disease of a non-PBC etiology
* Evidence of clinically significant hepatic decompensation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Absolute change in plasma ALP from Baseline to Week 12 | 12 weeks

SECONDARY OUTCOMES:
Percentage change in bilirubin, ALT, AST, and GGT from Baseline to Week 12 and Week 24 | 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Rossi, PharmD, Study Director — NGM Biopharmaceuticals, Inc
Locations (17):
- United States (6):
  - NGM Clinical Study Site 103, Phoenix, Arizona
  - NGM Clinical Study Site 108, Coronado, California
  - NGM Clinical Study Site 101, Detroit, Michigan
  - NGM Clinical Study Site 105, Durham, North Carolina
  - NGM Clinical Study Site 102, Dallas, Texas
  - NGM Clinical Study Site 113, San Antonio, Texas
- Australia (9):
  - NGM Clinical Study Site 602, Sydney, New South Wales
  - NGM Clinical Study Site 606, Sydney, New South Wales
  - NGM Clinical Study Site 609, Sydney, New South Wales
  - NGM Clinical Study Site 611, Sydney, New South Wales
  - NGM Clinical Study Site 614, Brisbane, Queensland
  - NGM Clinical Study Site 607, Adelaide, South Australia
  - NGM Clinical Study Site 608, Adelaide, South Australia
  - NGM Clinical Study Site 601, Melbourne, Victoria
  - NGM Clinical Study Site 613, Melbourne, Victoria
- New Zealand (2):
  - NGM Clinical Study Site 401, Auckland
  - NGM Clinical Study Site 402, Christchurch

REFERENCES:
- See also: Related Info — http://ngmbio.com/